CLINICAL TRIAL: NCT04786756
Title: Comparison of Ultrasound-Guided Lateral and Medial Approaches to Costoclavicular Brachial Plexus Block in Pediatric Patients Undergoing Unilateral Upper Exremity Surgery: A Randomized Controlled Double-Blinded Study
Brief Title: Comparison of Lateral and Medial Approaches to Costoclavicular Brachial Plexus Block in Pediatrics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Meltem Savran Karadeniz, Associate Professor, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Screening
Other Study IDs: 2019/1556
Record Dates: First submitted 2021-03-05; First posted 2021-03-08 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2022-01

CONDITIONS: Anesthesia, Local; Postoperative Pain
Keywords: Postoperative Analgesia; Upper Extremity Surgery; Costoclavicular Block; Brachial Plexus Block; Ultrasound Guidance
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine

STUDY DESIGN:
Intervention Model Description: RANDOMISED DOUBLE BLINDED INTERVENTIONAL
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lateral Approach of Costoclavicular Block (Active Comparator): US-guided lateral approach costoclavicular block with 1 mg/kg Bupivacaine (%0,25)
  Interventions: Drug: Bupivacaine 0.25% Injectable Solution
- Medial Approach of Costoclavicular Block (Active Comparator): US-guided medial approach costoclavicular block with 1 mg/kg Bupivacaine (%0,25)
  Interventions: Drug: Bupivacaine 0.25% Injectable Solution

INTERVENTIONS:
Drug: Bupivacaine 0.25% Injectable Solution — 1 mg/kg Bupivacaine (0.25%)
  Other Names: Marcaine

SUMMARY:
In upper extremity surgeries, the brachial plexus block can be performed with different techniques at various levels depending on the proximal and distal level of the surgery. In this study, we aim to compare the different approaches of US guided costoclavicular technique. Lateral approache is more common for the costoclavicular block area. However, more needle maneuvers are needed especially in pediatric patients because of the coracoid process. Medial approach is recommended to overcome this problem. Thus demonstrate the safety of upper extremity blocks, which is an important part of multimodal analgesia, and to determine the most ideal technique in the pediatric patient group who will undergo upper extremity surgery.

During the block application, the US imaging time, the difficulty level of needle imaging, the number of maneuvers required to reach the target image, whether additional maneuvers are required according to the local anesthetic distribution, the success of the block and the duration of the surgery, the total application time of the block and the duration of general anesthesia will be recorded. Mean arterial pressure and heart rate will be recorded at 30-minute intervals during the surgery. Standardized for pediatric patients The FLACC and Wong-Baker pain scores will be followed first 24 hours after surgery. The patient will be examined for motor and sensation, and analgesic doses will be recorded if used. Time to first pain identification, duration of sleep, patient and surgeon satisfaction will be recorded.

DETAILED DESCRIPTION:
Peripheral nerve blocks; It is widely used in daily practice for anesthesia or as a part of multimodal analgesia in most surgical procedures. In upper extremity surgeries, the brachial plexus block can be performed with different techniques at various levels depending on the proximal and distal level of the surgery. In this study, the aim is to compare postoperative analgesic effects of these two ultrasound-guided techniques in pediatric patients. In this study, we aim to compare the different approaches of US guided costoclavicular technique. Lateral approache is more common for the costoclavicular block area. However, more needle maneuvers are needed especially in pediatric patients because of the coracoid process. Medial approach is recommended to overcome this problem. Thus demonstrate the safety of upper extremity blocks, which is an important part of multimodal analgesia, and to determine the most ideal technique in the pediatric patient group who will undergo upper extremity surgery.

During the block application, the US imaging time, the difficulty level of needle imaging, the number of maneuvers required to reach the target image, whether additional maneuvers are required according to the local anesthetic distribution, the success of the block and the duration of the surgery, the total application time of the block and the duration of general anesthesia will be recorded. Mean arterial pressure and heart rate will be recorded at 30-minute intervals during the surgery. Standardized for pediatric patients The FLACC and Wong-Baker pain scores will be followed first 24 hours after surgery. The patient will be examined for motor and sensation, and analgesic doses will be recorded if used. Time to first pain identification, duration of sleep, patient and surgeon satisfaction will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing unilateral upper extremity surgery (distal midhumerus).
* ASA(American Society of Anesthesiology) 1-3
* Receiving family consent from the parents that they accept regional analgesia

Exclusion Criteria:

- Parents refusal

* Infection on the local anesthetic application area
* Infection in the central nervous system
* Coagulopathy
* Brain tumors
* Known allergy against local anesthetics
* Anatomical difficulties
* Syndromic patient

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 55 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-12-25 (Actual); Study Completion 2021-12-27 (Actual)

PRIMARY OUTCOMES:
Number of needle maneuvers | Up to 15 minutes
  Number of needle maneuvers according to local anesthetic distribution

SECONDARY OUTCOMES:
Ideal USG guided brachial plexus cords visualization/needle pathway planning time | Up to 15 minutes
  Practitioner's ideal image acquisition time
Needle tip and shaft imaging visualization | Up to 15 minutes
  Likert scale: 1-5
Requirement of additional needle maneuver due to insufficient local anesthetic distribution | Up to 15 minutes
  Extra needle redirection to cover neural tissue
Total procedure difficulty according to the anesthesiologist | Up to 15 minutes
  Likert Scale 1-5 (1:very hard 5:very easy)
Patient number requiring rescue analgesics | Intraoperative 2-4 hours
  If a ≥ 20% increase above preinduction values in MAP or HR was observed during the perioperative period, additional fentanyl dose (1 μg/kg) was applied intravenously.
Face, Legs Activity, Cry, Consolability (FLACC) scores | Up to 24 hours
  It corporates five categories of behavior, each scored on 0-2 point scale so that total score ranges from 0 to 10. Total scores of 0-3 is defined as mild or no pain, 4-7 as moderate, and 8-10 as severe pain.
Wong Baker FACES scale | Up to 24 hours
  The scale shows a series of faces ranging from a happy face at 0, or "no hurt", to a crying face at 10, which represents "hurts like the worst pain imaginable"
Motor blockade physical examination | Up to 24 hours
  Each nerve scored on 0-2 point scale so that total score ranges from 0 to 8. Total scores of 0 point is defined as absent motor blockade (full movement); 1 point as partial blockade (able to free movement only) or 2 point as complete blockade (unable to move). (Separately for these four nerves; N. Medianus, N. ulnaris, N. radialis and N. musculocutaneous).
Sensorial blockade physical examination | Up to 24 hours
  Each nerve scored on 0-2 point scale with pinprick test so that total score ranges from 0 to 8. Total scores of 0 point is defined as absent sensorial blockade (feels pain), 1 point as partial blockade (feels touch) or 2 point as complete blockade (no sense). (Separately for these four nerves; N. Medianus, N. ulnaris, N. radialis and N. musculocutaneous).
Time to first pain | Up to 24 hours
  Time to first analgesic
Patient number requiring additional analgesix | Up to 24 hours
  Number of patients who require IV morphine (0.03 mg/kg) and paracetamol (15 mg/kg)
Sleeping duration | Up to 24 hours
  Total hours of sleep first day
Complications/side effects | Up to 24 hours
  Possible complications related to costoclavicular block (such as vascular puncture, hematoma, pneumothorax, diaphragma palsy...)
Family satisfaction | Up to 24 hours
  Satisfaction score: 0: very unsatisfied 3: very satisfied
Surgeon satisfaction | Up to 24 hours
  Satisfaction score: 0: very unsatisfied, 3: very satisfied

CONTACTS AND LOCATIONS:
Overall Officials: Meltem Savran Karadeniz, Assoc.Prof., Principal Investigator — Istanbul University
Locations (1):
- Istanbul University, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Songthamwat B, Karmakar MK, Li JW, Samy W, Mok LYH. Ultrasound-Guided Infraclavicular Brachial Plexus Block: Prospective Randomized Comparison of the Lateral Sagittal and Costoclavicular Approach. Reg Anesth Pain Med. 2018 Nov;43(8):825-831. doi: 10.1097/AAP.0000000000000822. PMID 29923950